CLINICAL TRIAL: NCT02868645
Title: Interest of Serum Periostin Dosage in Patients With Bone Fibrous Dysplasia
Acronym: PERIOSTINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL15_0336
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Bone Fibrous Dysplasia
MeSH Terms: conditions — Fibrous Dysplasia of Bone | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with bone fibrous dysplasia (Experimental): Patients with bone fibrous dysplasia will have a blood sampling to assess periostin rate in serum
  Interventions: Biological: Blood sampling
- Control subjects (No Intervention): Control subjects will have no intervention

INTERVENTIONS:
Biological: Blood sampling — Patients with bone fibrous dysplasia will have blood sampling to assess periostin rate in serum
  Arms: Patients with bone fibrous dysplasia

SUMMARY:
Fibrous dysplasia is a rare bone disease which can cause pain and fractures. It has been shown that periostin is over expressed in fibrous component in patients bones ; but periostin has never been measured out in serum of patients, although it is easy to assess. This study aims to show whether serum periostin is elevated in serum of patients with fibrous dysplasia, and if it is more elevated in patients with severe forms of the disease.

ELIGIBILITY:
Inclusion Criteria:

* patients with fibrous dysplasia of the bone
* access to social security
* informed consent

Exclusion Criteria:

* no informed consent
* pregnancy
* patients with a history of conditions known to increase periostin serum (stade IV cancer, severe asthma, pulmonary fibrosis…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Periostin rate in serum | At inclusion

SECONDARY OUTCOMES:
Periostin rate in serum according to the number of fibrotic bones | At inclusion
Periostin rate in serum in patients with severe phenotype of the disease | At inclusion
Periostin rate in serum in patients with Mac Cune Albright syndrome | At inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Service de rhumatologie Pavillon F - Hôpital Edouard Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guerin Lemaire H, Merle B, Borel O, Gensburger D, Chapurlat R. Serum periostin levels and severity of fibrous dysplasia of bone. Bone. 2019 Apr;121:68-71. doi: 10.1016/j.bone.2019.01.004. Epub 2019 Jan 4. PMID 30616028